CLINICAL TRIAL: NCT04158154
Title: Transforming Hypertension Treatment in Nigeria Using a Type II Hybrid, Interrupted Time Series Design
Acronym: HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Abuja Teaching Hospital (Other); Resolve to Save Lives (Other)
Responsible Party: Principal Investigator, Mark Huffman, Professor of Medicine and Global Health Center Co-Director, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UATH/HREC/PR/2019/002; 1R01HL144708-01 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
Keywords: Hypertension; Nigeria; Primary Health Center
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This study applies an interrupted time series design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Health Care Centers (Experimental): Selected primary health care centers in Abuja will implement a culturally- and contextually-adapted intervention package based on the Kaiser Permanente Northern California and World Health Organization HEARTS programs for hypertension diagnosis and treatment.
  Interventions: Other: Evidence-based fixed-dose combination protocol based treatment

INTERVENTIONS:
Other: Evidence-based fixed-dose combination protocol based treatment — The intervention has been adapted based on a local needs' assessment including exploration of health care workers and patient's knowledge, attitudes, and behaviors related to HTN, causes, consequences, and treatment. Implementation pathways have been developed with particular attention to overcoming modifiable barriers to HTN treatment and control across capability, intentional, and system domains using CFIR. Sites will randomly be assigned to receive either: Step 1 amlodipine 5mg; Step 2 amlodipine 5 mg + losartan 50 mg (as 2 separate pills); Step 3 amlodipine 10 mg + losartan 100 mg (as 4 separate pills); Step 4 amlodipine 10/losartan 100/HCTZ 25 (as 2 single pill combo) or Step 1 amlodipine 5mg; Step 2 amlodipine 5 mg + losartan 50 mg (as 1 single pill combo); Step 3 amlodipine 10 mg + losartan 100 mg (as 2 single pill combo); Step 4 amlodipine 10/losartan 100/HCTZ 25 (as 2 single pill combo).

SUMMARY:
The purpose of the Transforming Hypertension Treatment in Nigeria Program is to improve awareness, treatment, and control of hypertension in Nigeria through the adaptation, implementation, and evaluation of the effectiveness and implementation of a system-level hypertension control program.

DETAILED DESCRIPTION:
This study includes the implementation and evaluation of a culturally- and contextually-adapted intervention package based on the Kaiser Permanente Northern California and World Health Organization HEARTS programs for hypertension diagnosis and treatment at primary health centers in Abuja, Nigeria. The intervention has been adapted based on a local needs' assessment including evidence synthesis and specific exploration of health care workers' knowledge, attitudes, and behaviors related to hypertension, causes, consequences, and treatment, including fixed-dose combination and patient self-management, and patients' knowledge, attitudes, and behaviors related to hypertension, causes, consequences, and treatment. Implementation pathways have been developed with particular attention to overcoming modifiable system- and patient-level barriers to hypertension treatment and control across capability, intentional, and system domains using the Consolidated Framework for Implementation Research. Preparedness and capacity have been assessed at primary health centers (e.g. available staff; information systems; use of clinical guidelines) through an adapted Service Availability and Readiness Assessment (SARA) instrument during the formative work for this study. The multi-level implementation package includes: 1) patient registration and empanelment (health system level), 2) standard treatment protocol (national policy level), 3) encouragement of fixed-dose combination therapy (health system level), 4) team-based care (health worker level), and 5) home blood pressure monitoring and health coaching (patient-level).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Elevated blood pressure (Systolic Blood Pressure ≥ 130 mmHg or Diastolic Blood Pressure ≥ 80 mmHg) documented or measured by a health care professional (e.g., physician, Community Health Extension Worker, or Community Health Officer).

Exclusion Criteria:

* Individuals who are not yet adults (minors)
* Prisoners or other detained individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21922 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Slope of Treatment Rate | Through study completion, 45 months
  Hypertension treatment using any blood pressure lowering drug. Treatments rates are calculated monthly, over 9 months of baseline and 39 months of intervention.
Change from Baseline Slope of Control Rate | Through study completion, 45 months
  Hypertension control is defined as a Systolic Blood Pressure <140 mmHg and Diastolic Blood Pressure <90 mmHg. Control rates are calculated monthly, over 9 months of baseline and 39 months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Huffman, MD, MPH, Principal Investigator — Northwestern University Feinberg School of Medicine; Dike B Ojji, MD, PhD, Principal Investigator — University of Abuja Teaching Hospital
Locations (60):
- Nigeria (60):
  - Agyana PHC, Abaji, Abaji
  - Central PHC, Abaji, Abaji
  - Gawu PHC, Abaji, Abaji
  - Low Cost PHC, Abaji, Abaji
  - Naharati PHC, Abaji, Abaji
  - New Township Clinic, Abaji, Abaji
  - Rimba PHC, Abaji, Abaji
  - Yaba PHC, Abaji, Abaji
  - Dakwa PHC, Abuja, Abuja Municipal Area Council
  - Gbagarape PHC, Abuja, Abuja Municipal Area Council
  - Gidan Mangoro PHC, Abuja, Abuja Municipal Area Council
  - Gosa PHC, Abuja, Abuja Municipal Area Council
  - Gwagwa PHC, Abuja, Abuja Municipal Area Council
  - Jikwoyi PHC, Abuja, Abuja Municipal Area Council
  - Kagini PHC, Abuja, Abuja Municipal Area Council
  - Karon Majigi PHC, Abuja, Abuja Municipal Area Council
  - Karshi PHC, Abuja, Abuja Municipal Area Council
  - Karu PHC, Abuja, Abuja Municipal Area Council
  - Kuchingoro PHC, Abuja, Abuja Municipal Area Council
  - Lugbe PHC, Abuja, Abuja Municipal Area Council
  - New Garki Apo PHC, Abuja, Abuja Municipal Area Council
  - Orozo PHC, Abuja, Abuja Municipal Area Council
  - Pykassa PHC, Abuja, Abuja Municipal Area Council
  - Byazhin PHC, Bwari, Bwari
  - Dei-Dei PHC, Bwari, Bwari
  - Kawu PHC, Bwari, Bwari
  - Kogo PHC, Bwari, Bwari
  - Mpape PHC, Bwari, Bwari
  - Sabon Gari PHC, Bwari, Bwari
  - Shere PHC, Bwari, Bwari
  - Ushafa PHC, Bwari, Bwari
  - Anagada PHC, Gwagwalada, Gwagwalada
  - Dagiri CPHC, Gwagwalada, Gwagwalada
  - Dobi PHC, Gwagwalada, Gwagwalada
  - Dukpa PHC, Gwagwalada, Gwagwalada
  - Gwagwalada Township Clinic, Gwagwalada, Gwagwalada
  - Gwako PHC, Gwagwalada, Gwagwalada
  - Old-Kutunku PHC, Gwagwalada, Gwagwalada
  - Paikon PHC, Gwagwalada, Gwagwalada
  - Rafin Zurfi PHC, Gwagwalada, Gwagwalada
  - Yimi PHC, Gwagwalada, Gwagwalada
  - Zuba PHC, Gwagwalada, Gwagwalada
  - Chukuku PHC, Kuje, Kuje
  - Gaube CPHC, Kuje, Kuje
  - Gudunkarya PHC, Kuje, Kuje
  - Gwargada PHC, Kuje, Kuje
  - Kiyi PHC, Kuje, Kuje
  - Kuje PHC, Kuje, Kuje
  - Kujekwa PHC, Kuje, Kuje
  - Pegi PHC, Kuje, Kuje
  - Ashara PHC, Kwali, Kwali
  - Dabi Bako CPHC, Kwali, Kwali
  - Dafa PHC, Kwali, Kwali
  - Gomani PHC, Kwali, Kwali
  - Kwaita Hausa PHC, Kwali, Kwali
  - Kwaita Model PHC, Kwali, Kwali
  - Kwali PHC, Kwali, Kwali
  - Petti PHC, Kwali, Kwali
  - Wako PHC, Kwali, Kwali
  - Yangoji PHC, Kwali, Kwali

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared through NHLBI BioLINCC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion.
Access Criteria: Access to study data will be managed through NHLBI BioLINCC.

REFERENCES:
- [Derived] Ye J, Hirschhorn LR, Baldridge AS, Jamro EL, Orji IA, Shedul GL, Ripiye NR, Ojo TM, Eze H, Shedul GJ, Ugwuneji EN, Okoli RCB, Ale BM, Osagie S, Sanuade OA, Iyer G, Kandula NR, Ojji DB, Huffman MD. Implementation outcomes from the Hypertension Treatment in Nigeria program: results from a type 2 hybrid interrupted time series trial. Implement Sci. 2025 Nov 26;21(1):1. doi: 10.1186/s13012-025-01472-1. PMID 41299526
- [Derived] Baldridge AS, Odukwe A, Dabiri O, Mobisson LN, Munnee MM, Ogboye A, Aryee DNK, Mwale R, Akpakli J, Orji IA, Okoli RCB, Ripiye NR, Ojji DB, Huffman MD, Kandula NR, Hirschhorn LR. Implementation of the Extension for Community Healthcare Outcomes Model for Hypertension Education of Frontline Health Care Workers in the Federal Capital Territory, Nigeria: Explanatory Sequential Mixed Methods Evaluation. J Med Internet Res. 2025 Apr 24;27:e66351. doi: 10.2196/66351. PMID 40273438
- [Derived] Shedul GL, Ripiye N, Jamro EL, Orji IA, Shedul GJ, Ugwuneji EN, Okpetu E, Ale BM, Osagie S, Baldridge AS, Kandula NR, Huffman MD, Ojji D, Hirschhorn L. Supportive supervision visits in a large community hypertension programme in Nigeria: implementation methods and outcomes. BMJ Open Qual. 2025 Mar 24;14(1):e003163. doi: 10.1136/bmjoq-2024-003163. PMID 40127954
- [Derived] Baldridge AS, Orji IA, Shedul GL, Iyer G, Jamro EL, Ye J, Akor BO, Okpetu E, Osagie S, Odukwe A, Dabiri HO, Mobisson LN, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Enhancing hypertension education of community health extension workers in Nigeria's federal capital territory: the impact of the extension for community healthcare outcomes model on primary care, a quasi-experimental study. BMC Prim Care. 2024 Sep 7;25(1):334. doi: 10.1186/s12875-024-02579-y. PMID 39244554
- [Derived] Baldridge AS, Goldstar N, Bellinger GC, DeNoma AT, Orji IA, Shedul GL, Okoli RCB, Ripiye NR, Odukwe A, Dabiri O, Mobisson LN, Ojji DB, Huffman MD, Kandula NR, Hirschhorn LR. Formative Evaluation and Adaptation of a Hypertension Extension for Community Health Outcomes Program for Healthcare Workers within the Federal Capital Territory, Nigeria. Glob Heart. 2023 Nov 27;18(1):64. doi: 10.5334/gh.1277. eCollection 2023. PMID 38045112
- [Derived] Ojji DB, Sancilio A, Shedul GL, Orji IA, Chopra A, Abu J, Akor B, Ripiye N, Akinlade F, Okoye D, Okpetu E, Eze H, Odoh E, Baldridge AS, Tripathi P, Abubakar H, Jamda AM, Hirschhorn LR, McDade T, Huffman MD. Nigeria healthcare worker SARS-CoV-2 serology study: Results from a prospective, longitudinal cohort. PLOS Glob Public Health. 2023 Jan 17;3(1):e0000549. doi: 10.1371/journal.pgph.0000549. eCollection 2023. PMID 36962953
- [Derived] Sanuade OA, Ale BM, Baldridge AS, Orji IA, Shedul GL, Ojo TM, Shedul G, Ugwuneji EN, Egenti N, Omitiran K, Okoli R, Eze H, Nwankwo A, Hirschhorn LR, Chopra A, Ye J, Tripathi P, Banigbe B, Kandula NR, Huffman MD, Ojji DB; Hypertension Treatment in Nigeria Program Investigators. Fixed-dose combination therapy-based protocol compared with free pill combination protocol: Results of a cluster randomized trial. J Clin Hypertens (Greenwich). 2023 Feb;25(2):127-136. doi: 10.1111/jch.14632. Epub 2023 Jan 20. PMID 36660886
- [Derived] Baldridge AS, Aluka-Omitiran K, Orji IA, Shedul GL, Ojo TM, Eze H, Shedul G, Ugwuneji EN, Egenti NB, Okoli RCB, Ale BM, Nwankwo A, Osagie S, Ye J, Chopra A, Sanuade OA, Tripathi P, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Hypertension Treatment in Nigeria (HTN) Program: rationale and design for a type 2 hybrid, effectiveness, and implementation interrupted time series trial. Implement Sci Commun. 2022 Aug 2;3(1):84. doi: 10.1186/s43058-022-00328-9. PMID 35918703
- [Derived] Ojji DB, Baldridge AS, Orji IA, Shedul GL, Ojo TM, Ye J, Chopra A, Ale BM, Shedul G, Ugwuneji EN, Egenti NB, Aluka-Omitiran K, Okoli RCB, Eze H, Nwankwo A, Banigbe B, Tripathi P, Kandula NR, Hirschhorn LR, Huffman MD; Hypertension Treatment in Nigeria Program Investigators. Characteristics, treatment, and control of hypertension in public primary healthcare centers in Nigeria: baseline results from the Hypertension Treatment in Nigeria Program. J Hypertens. 2022 May 1;40(5):888-896. doi: 10.1097/HJH.0000000000003089. Epub 2022 Jan 15. PMID 35034080